CLINICAL TRIAL: NCT02315248
Title: Salivary-based Bone Loss Marker Detection Platform for Point-of-care Screening - Phase II Study
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2014-0108
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2014-12

CONDITIONS: Osteoporosis
Keywords: bone density
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Salivary biosamples will be stored for assaying osteocalcin (OC) and deoxypyridinoline (DPD) levels
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Quantitative computed tomography scan for bone density analysis — A low radiation dose quantitative computed tomography (QCT) of the spine (L1 and L2) and the hips will be performed to measure bone density in the spine and hips.

SUMMARY:
The purpose of this study is to validate a human saliva sample analyzer technique designed to screen for low bone density and osteoporosis. The analyzer technique is meant to be a simple, noninvasive, easy-to-use, cost-effective, and routine means of diagnosing bone turnover using a point-of-care device that monitors salivary markers of bone turnover in a screening patient population that is at risk for low bone density or osteoporosis.

DETAILED DESCRIPTION:
Primary objective: To validate the performance of human saliva sample analyzer LFA technique against bone density as measured by quantitative computed tomography (QCT).

Secondary objective: To validate the performance of human saliva sample analyzer LFA technique against salivary ELISA method (gold standard).

Number of sites: Single site at the University of Mississippi Medical Center

The purpose of this prospective Phase II observational study is to further refine a proprietary device and test it in a screening population composed of women 50 years of age or older who are at risk for low bone density or osteoporosis (N=200). After screening for inclusion and exclusion criteria and obtaining informed consent, participants will provide a salivary sample and will undergo quantitative computed tomography (QCT) at the same visit (Visit 1, Day 0). No additional visits are planned. Bone mineral density (BMD) will be measured by diagnostic radiologists using QCT techniques and serve as the gold standard for the study. Salivary samples will be analyzed by a lab at UMMC for concentrations of osteocalcin (OC) and deoxypyridinoline (DPD) using enzyme-linked immunosorbent assay (ELISA) techniques, while blinded to BMD measurements. De-identified and coded salivary sample will be shipped to IOS who will measure concentrations of OC and DPD using lateral flow assay (LFA), while blinded to BMD measurements.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥50 years of age and referred for standard of care screening mammogram.
* Ability to provide salivary samples.
* Ability to lie flat on the CT scanner.
* Ability and willingness to provide signed and dated informed consent.

Exclusion Criteria:

* Any known bone metabolism disorder (other than osteoporosis or low bone density) including sickle cell disease, current neoplastic disease, metastatic disease or any neoplastic disease involving the bones (including leukemia), or Paget's disease.
* Body weight exceeds the weight limit (>400lbs) of the CT table.
* Vulnerable subjects including pregnant women and prisoners.
* Subjects who have had prior QCT imaging to measure bone density.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of asymptomatic women 50 years of age or older who present for a screening mammogram and are at risk for low bone density or osteoporosis (N=200).
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Validation of human saliva sample analyzer LFA technique against measured bone density | 20 months
  To validate the performance of human saliva sample analyzer LFA technique against bone density as measured by quantitative computed tomography (QCT).

SECONDARY OUTCOMES:
Validation of human saliva sample analyzer LFA technique against ELISA (gold standard) | 20 months
  To validate the performance of human saliva sample analyzer LFA technique against salivary ELISA method (gold standard).

CONTACTS AND LOCATIONS:
Overall Officials: Manal Bashay, MS, Principal Investigator — Intelligent Optical Systems Inc.
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States